CLINICAL TRIAL: NCT06969859
Title: Multicentre Randomised Controlled Trial of Pulsed Electro-Magnetic Field Therapy for Treatment of Midportion Achilles Tendinopathy（EM-MAT Trial)
Brief Title: Pulsed Electro-Magnetic Field Therapy for Treatment of Midportion Achilles Tendinopathy
Acronym: EM-MAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor of Orthopaedics and Traumatology, CUHK Head of the Foot and Ankle Team / Honorary Associate Consultant, Prince of Wales Hospital Specialist in Orthopaedics and Traumatology, CUHK Medical Centre, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025.193
Record Dates: First submitted 2025-04-24; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Mid-portion Achilles Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEMF Therapy + Exercise (Experimental)
  Interventions: Device: PEMF; Behavioral: Alfredson eccentric training program
- sham Therapy + Exercise (Sham Comparator)
  Interventions: Behavioral: Alfredson eccentric training program

INTERVENTIONS:
Device: PEMF — The PEMF will be delivered using a BIXEPS device (Quantum Tx, Singapore) ; It is utilised by the patient placing the leg into the machine. This device is operated by participant individualized NFC cards, which will be centrally programmed to deliver either active PEMF (uniform 1mT, 50Hz) or sham PEMF (0mT, 0Hz) for 30 minutes. Because this biophysical intervention is non-invasive, and the electromagnetic fields emitted into the legs do not generate any sensation (e.g. heat, sound), participants will be blinded to the treatment. The protocol will be 180 minutes of PEMF therapy, performed in six 30-minute sessions 3 times a week and completed in 2 weeks.
  Arms: PEMF Therapy + Exercise
Behavioral: Alfredson eccentric training program — All participants will be subject to a standardised rehabilitation exercise region consisting of stretching and eccentric exercises following the Alfredson protocol. The 12-week program will be taught by a physiotherapist or athletic trainer and supplemented by video tutorials. The regime begins with three 30-second static stretches for the gastrocnemius (knee extension) and soleus (knee flexion) muscles with 1-minute rest between each stretch. The 2nd part is eccentric exercises to the calves following the Alfredson protocol. This will be three sets of eccentric exercises lasting 12 weeks, with 15 sets twice a day. If participants are unable to complete three sets of 15 repetitions, they can start with fewer repetitions and sets (at least 2 sets of 10 repetitions each) and gradually increase to the total number of sets. Participants will perform the static stretching exercises from Step 1 at the end of each session

SUMMARY:
This is a multi-centre, randomised, double-blind, placebo-controlled trial with two parallel groups in a 1:1 allocation to study the efficacy of Pulsed Electromagnetic Field Therapy (PEMF) in patients with mid-portion Achilles tendinopathy. All participants will be randomly divided into two groups: an intervention group (active PEMF and standard rehabilitation exercise) and a control group (sham PEMF and standard rehabilitation exercise). All self-reported, functional, and ultrasound findings will be evaluated by the investigator at baseline assessment, 1-month, 2-month, 3-month, 6-month and 12-month follow-up after initiating the intervention.

The researcher will obtain written consent from all participants before the start of this study. All eligible participants will be informed about this study and given enough time to consider whether or not to participate; the clinician/research staff will answer all questions asked by the participants. The trial will be conducted in accordance with the Declaration of Helsinki and the ICH-GCP. Clinical research ethics approval for the trial will be obtained from the Joint Clinical Research Ethics Committee of The Chinese University of Hong Kong. All participants will be recruited from the clinics and centres of the participating institutions.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age)
* Clinical diagnosis of mid-Achilles tendinopathy
* VISA-A score of <60
* Ultrasound evidence of Achilles tendinopathy (thickening >7mm)

Exclusion Criteria:

* Previous invasive treatment to the Achilles tendon (e.g. rupture repair, PRP injection etc)
* Contraindication to PEMF (e.g. pregnancy, pacemakers)
* Physical or psychological comorbidities impairing the ability to complete assessments (eg neurological deficits etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sports Assessment (VISA-A) | Baseline;2-month;3-month;6-month;12month follow-up after initiating the intervention
  The primary outcome measure will be the Victorian Institute of Sport Assessment (VISA-A) questionnaire, available in either the original English or validated Chinese version, depending on the participant's native language. This specific scoring system developed for the Achilles tendon is the most widely used score for clinical Achilles research. The VISA-A is scored on a scale of 0 to 100; lower scores indicate more severity of symptoms, while a score of 100 indicates a healthy and pain-free Achilles tendon.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline;2-month;3-month;6-month;12month follow-up after initiating the intervention
  Numeric Pain Rating Scale (NPRS) is a pain screening tool, commonly used to assess pain severity using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable
Foot and Ankle Outcome Scores (FAOS) | Baseline;2-month;3-month;6-month;12month follow-up after initiating the intervention
  The FAOS is a validated patient-reported scoring system used for general foot and ankle problems. It is split into five categories: symptoms, pain, daily activities, sporting function, and quality of life. Scores range from 0 to 100, with 100 denoting no problems and 0 denoting severe problems.
Achilles tendon resting angle (ATRA) | Baseline;2-month;3-month;6-month;12month follow-up after initiating the intervention
  The ATRA will measure participants' tendon length/tension. Participants should be positioned in a prone position with the knee flexed to 90 degrees. The assessor will use a dynamic joint goniometer to measure the angle at which the foot passively falls.
Tendon thickness | Baseline;2-month;3-month;6-month;12month follow-up after initiating the intervention
  Using B-mode ultrasound scanning, the probe is moved from the medial to the lateral aspect of the Achilles tendon until a planar image of the Achilles tendon is clearly shown. The probe was adjusted straight perpendicular to the tendon fibres. A greyscale sonogram is acquired, and the tendon thickness is measured using the maximum thickness. Less than 5.3 mm was considered a healthy value for the Achilles tendon.
Tendon cross sectional area | Baseline;2-month;3-month;6-month;12month follow-up after initiating the intervention
  The cross-sectional area will be measured using B mode. After identifying the region of interest (the thickest portion or pathological site) in the longitudinal view, the transducer is rotated 90° to switch to the short-axis view (axial ultrasound view, as shown in the figure) for cross-sectional measurement. The cross-sectional area (CSA) is then recorded.
Tendon vascularity | Baseline;2-month;3-month;6-month;12month follow-up after initiating the intervention
  Vascularity will be documented using the Ohberg score. Using the Doppler mode on the ultrasound machine, the transducer is placed vertically to obtain a sagittal view of the softest area of the Achilles tendon. Pressure on the skin from the transducer should be kept to a minimum to prevent occlusion of blood vessels. The colour box is focused on the dorsal aspect of the tendon. The assessor will spend one minute exploring the blood flow over the tendon to find the area of maximum Doppler flow. After locating the area, sonograms are taken to determine the Öhberg score. Higher scores indicate more Doppler blood flow in the peritendinous and intratendinous tissues. Healthy tendons (Ohberg score of 0) have no blood vessels in the Achilles tendon.
Tendon elasticity | Baseline;2-month;3-month;6-month;12month follow-up after initiating the intervention
  Shear wave elastography (SWE) can be used to quantify soft tissue stiffness. Once the optimal scan plane of the tendon is determined, the SWE function is activated. It enters penetration mode and the measured stiffness range is normalized to 0-600 kPa. The SWE color card (H × W: 1.4 cm × 1.3 cm) is placed immediately above the upper edge of the calcaneus. After the color signal stabilized for five seconds, the electrogram was recorded and stored. Tendon stiffness was measured using a Q-box stiffness meter. Depending on the size of the tendon, the diameter of the circular measuring area (Q-box) is set to 2 mm, which covers the Achilles tendon and excludes other adjacent soft tissues. The Q-box is located in the center of the tendon on the SWE color map. For each Q-box, the average tendon stiffness (in kPa) is measured.
Calf muscle strength | Baseline;2-month;3-month;6-month;12month follow-up after initiating the intervention
  The hand-held dynamometer will be used to quantify isometric muscle strength (in kilograms) during ankle dorsiflexion and plantarflexion. Participants will maintain a maximal voluntary isometric contraction for 3 seconds. Three trials will be performed for each movement, with 30-second rest intervals between trials to minimize fatigue.

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: From 2028-5-31 to 2033-5-28